CLINICAL TRIAL: NCT07080918
Title: EFFECTS OF IRRIGATION NEEDLES WITH DIFFERENT DESIGNS USED DURING ENDODONTIC TREATMENT ON POSTOPERATIVE PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Damla Kırıcı, Damla Kırıcı, Akdeniz University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 143
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Lower Molars With Irreversible Pulpitis
Keywords: root canal treatment, conventional needle irrigation, irrigation needle design, postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): For group 1, an open-ended notched irrigation needle (Endo-Top, Cerkamed, Stalowa Wola, Poland)Raito, China)
  Interventions: Procedure: Irrigation
- Group 2 (Experimental): For group 2, a closed-ended single orifice irrigation needle (Scope Endo Fx Ject, Turkey)
  Interventions: Procedure: Irrigation
- Group 3 (Experimental): For group 3,a closed-ended double orifice irrigation needle (Double Sideport, Raito, China)
  Interventions: Procedure: Irrigation

INTERVENTIONS:
Procedure: Irrigation — Irrigation procedures were performed with needles of different designs, each 30 G, for three different groups

SUMMARY:
This study is aimed to comparatively evaluate the effects of different irrigation needle designs used during endodontic treatment on postoperative pain and to provide information on which needle designs may be more advantageous in clinical applications based on the findings obtained.

DETAILED DESCRIPTION:
In this study, the mandibular molars of patients aged 18-65 who were diagnosed with symptomatic irreversible pulpitis and underwent root canal treatment at the Endodontics Clinic of Akdeniz University Faculty of Dentistry between January 2023 and January 2024 were included. Postoperative pain assessment forms obtained during the routine follow-up of the patients were included in the study.The study included patients who underwent routine root canal treatment procedures at the Endodontics clinic of Akdeniz University Faculty of Dentistry, where the treatments were performed by a single dentist. The age, gender, systemic diseases, root canal structure, periapical condition, irrigation needle design used during endodontic treatment, and pre- and post-treatment pain severity of the patients included in the study were obtained from patient records and follow-up forms.

Before the procedure, the patients' medical and dental histories were taken, and preoperative pain levels were recorded. Each patient received an inferior alveolar nerve block using a 2 ml local anesthetic solution (Ultracain D-S forte, Sanofi, France) containing 80 mg articaine hydrochloride and 0.024 mg epinephrine hydrochloride. After the teeth related to the rubber dam were isolated, caries and any existing restorations were removed using diamond burs, and a standard endodontic access cavity was prepared.

For canal length determination, #10 K-type (Perfect, China) hand files were used, and the working length was determined with an electronic apex locator (Woodpecker, Endo Radar Pro, China) and confirmed radiologically.

Root canal preparation was performed using an endodontic motor (Woodpecker, Endo Radar Pro, China) and a nickel-titanium rotary instrument system (Scope Endodontic System, Turkey) at a speed of 300 rpm and a torque of 2 N/cm. Apical preparation was completed to a size three larger. During shaping, at the point where apical resistance was encountered, excessive torsional loading was prevented by removing the files from the canal, cleaning the debris from the files, and irrigating the root canals.

During the shaping process, the root canals were rinsed with 2 ml of 2.5% NaOCl after each file change and recapitulated with a #10K file. After the root canal preparation procedure was completed, each canal was rinsed with 5 ml of 2.5% NaOCl, and the NaOCl solution was activated using an endoactivator in three 20-second cycles. 5 ml of distilled water was applied to remove NaOCl residues from the canal. Then, 2 ml of 17% EDTA (Endo-Solution, Cerkamed, Stalowa Wola, Poland) was applied for 1 minute. To neutralize the EDTA residues, each canal was finally irrigated with 5 ml of distilled water.

Irrigation procedures were performed with needles of different designs, each 30 G, for three different groups:

For group 1, an open-ended notched irrigation needle (Endo-Top, Cerkamed, Stalowa Wola, Poland) was used, For group 2, a closed-ended single orifice irrigation needle (Scope Endo Fx Ject, Turkey) was used, For group 3, a closed-ended double orifice irrigation needle (Double Sideport, Raito, China) was used.

The irrigation needles were used 2 mm shorter than the working length. The root canals were shaped using appropriate paper points (Meta Biomed, Korea). The root canals were filled using the lateral condensation technique with gutta-percha (Diadent Group International, Canada) and epoxy resin-based root canal paste (Dentac, Turkey). The permanent restoration was completed with light-curing composite (Coltene Whaledent Brilliant Ng, Switzerland), and occlusal adjustment was checked. Patients were prescribed 400 mg of ibuprofen and advised to use it when absolutely necessary.Evaluation of Postoperative Pain Patients were given a postoperative pain assessment form that included a visual analog scale (VAS) to evaluate their postoperative pain levels. Patients were informed about the topic and asked to record their pain levels and analgesic usage on the provided form at 6, 24, 48, 72 hours, and on the 7th day. Patients were called for a follow-up session one week later, and the given forms were collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients ranging between 18 and 65 years in age,
* Patients with preoperative pain score ranging from moderate to severe (4-10) on a visual analog scale (VAS, 0-10)
* Mandibular molar teeth were diagnosed with symptomatic irreversible pulpitis

Exclusion Criteria:

* Patients with systemic diseases,

  * Pregnancy or lactation
  * Teeth with periapical lesions,
  * Teeth that previous root canal treatment,
  * Teeth with calcified canals,
  * Teeth with periodontal diseases,
  * Teeth with sensitivite to percussion and palpation,
  * Teeth with bruxism/traumatic occlusion,
  * Teeth with crown or root fractures,
  * Teeth with internal or external resorption,
  * Teeth with immature/open apex,
  * Patients who had taken antibiotics in the last two weeks,
  * Patients who had taken analgesic or anti-inflammatory drugs within the last 12 hours,
  * Patients missing consent and follow-up forms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative pain with VAS after root canal treatment | 6, 24, 48, 72 hours, and on the 7th day

CONTACTS AND LOCATIONS:
Overall Officials: Damla Kırıcı, Associate Prof, Study Chair — Akdeniz University; Damla Kırıcı, ASSOCİATE PROF, Study Chair — AkdenizUniversity; DAMLA KIRICI, ASSOCİATE PROF, Study Chair — AKDENİZ UNİVERSİTY
Locations (1):
- AkdenizUniversity, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Yersel A, Kirici D. The effect of the design of the irrigation needle used during endodontic treatment on postoperative pain: a randomize clinical trial. Sci Rep. 2026 Jan 7;16(1):4452. doi: 10.1038/s41598-025-34420-6. PMID 41501119